CLINICAL TRIAL: NCT00872287
Title: Randomized Controlled Study of Different Pain Scores in Single Transumbilical Incision Laparoscopic Cholecystectomy Versus Classic Laparoscopic Cholecystectomy
Brief Title: Pain in Single Incision Laparoscopic Surgery Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Responsible Party: Evangelos C. Tsimoyiannis/G. Hatzikosta General Hospital, Ioannina, Greece, G. Hatzikosta General Hospital, Ioannina, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GH-1948-01; GHDS-12345-1
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: minimally invasive surgery; scarless cholecystectomy; new techniques in laparoscopy; invisible scar; single port access; abdominal pain; shoulder pain
MeSH Terms: conditions — Abdominal Pain; Shoulder Pain | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Cholecystectomy (Active Comparator): Four ports classic laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic Cholecystectomy
- SILS (Active Comparator): Single transumbilical incision laparoscopic cholecystectomy
  Interventions: Procedure: SILS

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Four ports classic laparoscopic cholecystectomy
  Arms: Laparoscopic Cholecystectomy
Procedure: SILS — Single transumbilical incision laparoscopic cholecystectomy
  Arms: SILS

SUMMARY:
The attempt to further reduce the operative trauma in laparoscopic cholecystectomy led in new techniques, as Natural Orifice Transluminal Endoscopic Surgery (NOTES) and Single Incision Laparoscopic Surgery (SILS). These new techniques are considered as painless procedures, but there are not any publications to study a possible different pain score in new techniques versus classic laparoscopic cholecystectomy. In this randomized controlled study the researchers have investigated the pain scores, the incidence of nausea and vomiting and analgesics request after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index less than 30
* Attacks of cholelithiasis

Exclusion Criteria:

* Body Mass Index more than 30
* Signs of acute cholecystitis

Ages: 28 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
SILS cholecystectomy, except the invisible scar, has significantly less abdominal and shoulder pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos C. Tsimoyiannis, M.D., Study Chair — G. Hatzikosta General Hospital, Ioannina, Greece
Locations (1):
- G. Hatzikosta General Hospital, Ioannina, Epirus, Greece

REFERENCES:
- [Derived] Tsimoyiannis EC, Tsimogiannis KE, Pappas-Gogos G, Farantos C, Benetatos N, Mavridou P, Manataki A. Different pain scores in single transumbilical incision laparoscopic cholecystectomy versus classic laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2010 Aug;24(8):1842-8. doi: 10.1007/s00464-010-0887-3. Epub 2010 Feb 20. PMID 20174950